CLINICAL TRIAL: NCT06565689
Title: A Multi-center, Open-Label, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of YK012 in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of YK012
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Excyte Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YK012-1
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YK012 (Experimental): Drug: YK012 Patients will be administered with YK012 by intravenous infusion every two weeks (Q2W, 4 weeks in a treatment cycle). Treatment will be continued until disease progression, intolerable toxicity, withdrawal of consent, patient being lost to follow-up, death or up to 6 cycles, whichever occurs first.
  Interventions: Drug: YK012

INTERVENTIONS:
Drug: YK012 — YK012 is a bispecific antibody targeting CD19 on B cells and CD3 on T cells leading to T cell-mediated cytotoxicity of malignant B cells
  Other Names: YK012 for Injection

SUMMARY:
This study aims to provide a basis for further clinical development of YK012.

DETAILED DESCRIPTION:
This study is the first-in-human clinical trial to evaluate the safety, tolerability, pharmacokinetic (PK) profile and preliminary efficacy of YK012 in patients with relapsed or refractory B-cell non-Hodgkin lymphoma (R/R B-NHL).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any study-related procedures, including screening visits.
2. Males or females aged ≥ 18 to ≤ 65 years.
3. Participants with an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 1.
4. Participants with an estimated survival time of more than 12 weeks.
5. Participants with relapsed or refractory B-NHL. These patients' disease history must meet the following World Health Organization (WHO) diagnostic subtypes of B-NHL : follicular lymphoma (FL), MALT lymphoma, lymphoplasmacytic lymphoma (LPL), mantle cell lymphoma (MCL), small lymphocytic lymphoma (SLL), diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), grey zone lymphoma, Burkitt lymphoma.
6. Participants have previously received rituximab Treatment (unless rituximab is intolerant) and at least second-line therapy.
7. Participants with at least one evaluable tumor lesion per the Lugano 2014 criteria, i.e., a lymph node lesion > 15 mm in long diameter or an extranodal lesion > 10 mm in long diameter according to computed tomography (CT) cross-sectional imaging.
8. Adverse reactions caused by previous treatment have recovered to below level 1 assessed by NCI CTCAE v5.0 before screening (except hair loss).
9. Participants with essentially normal function of hematology, liver, and kidney function.
10. Female participants of childbearing potential must have a negative blood pregnancy test and agree to use reliable methods of contraception (hormonal or barrier methods or sexual abstinence) with their partner throughout the study period and until 3 months after the last dose.
11. Male participants must agree to use reliable methods of contraception (barrier methods or sexual abstinence) and avoid sperm donation throughout the study period and until 90 days after the last dose.

Exclusion Criteria:

1. Participants who meet any of the following exclusion criteria will not be included in this study:

   Treatment with biologic targeted therapy or anti-tumor immunotherapy within 4 weeks prior to the first dose of YK012; Participants who have received chemotherapy within 4 weeks prior to the first dose of YK012; Participants who have received small molecule targeted agents within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of YK012; Participants who have received other investigational agents within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of YK012; Participants who have received radical/extensive radiotherapy within 4 weeks prior to the first dose of YK012, or local palliative radiotherapy within 2 weeks prior to the first dose of YK012, or acute toxicity induced by previous radiotherapy have not recovered to grade ≤1; Participants who have received autologous HSCT within 12 weeks prior to the first dose of YK012; Participants who have received allogeneic HSCT or organ transplant; Participants who have received chimeric antigen receptor T cell (CAR-T) immunotherapy.
2. History of malignancy other than B-cell NHL within 5 years prior to study entry, except for local cancers that have been clearly cured or have been free of disease for at least 5 consecutive years.
3. Participants with clinically symptomatic metastases to the central nervous system or meninges, or other evidence of uncontrolled metastases to the CNS or meninges, judged by the Investigator.
4. a) History of or current relevant CNS pathology as epilepsy, seizure, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis; b) Evidence for presence of inflammatory lesions and/or vasculitis on cerebral MRI.
5. Participants with a history or evidence of serious cardiovascular disease, including but not limited to:

   Acute coronary; Coronary angioplasty or stent implantation within 6 months prior to first dose of YK012; Clinically significant unstable arrhythmias (e.g., atrial fibrillation) , however, whose atrial fibrillation have been controlled for over 30 days prior to the first dose of YK012 were allowed to be enrolled; Severe cardiac rhythm abnormalities; Grade III or higher congestive heart failure as defined by the New York Heart Association (NYHA) standards; Cardiac valve morphological abnormalities recorded by ECHO (≥ grade 2), those participants with grade 1 cardiac valve morphological abnormalities (such as mild regurgitation/stenosis) were allowed to be enrolled, but participants with moderate valve thickening were excluded; Left ventricular ejection fraction (LVEF) below lower limit of the study center, or LVEF<50% if there is no lower limit at the research center; QTcF ≥ 470 msec (female) or ≥ 450 msec (male)； Implantable defibrillator; Participants with clinically uncontrollable hypertension (i.e., SBP≥160 mm Hg and/or DBP≥100 mm Hg).
6. Known allergy to monoclonal antibody drugs or immunoglobulin.
7. Participants who have undergone any major organ surgery or significant trauma within 4 weeks prior to the first dose of YK012, or those requiring elective surgeries during the study, and all AEs associated with surgery or significant trauma have not recovered before the first dose of the YK012.
8. Regular dose of systemic corticosteroids during the 4 weeks prior to initiation of study drug or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent during the trial, or any other systemic immunosuppressive therapy within 4 weeks prior to study entry.
9. The results of serological testing for the virus are clinically significant as judged by the investigator.
10. Participants with uncontrolled active infections currently require systemic anti-infective therapy, except for local treatment.
11. Participants with uncontrollable space effusion (e.g. pleural effusion, abdominal effusion, pericardial effusion, etc.), as judged by the Investigator.
12. Pregnant or lactating women.
13. Participants with mental disorders or poor protocol compliance.
14. Participants who have used live attenuated vaccines within 4 weeks prior to the first dose of YK012.
15. Participants with any other condition or circumstance that would, in the discretion of the Investigator, make the subject unsuitable for participation in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of subjects with adverse events (AEs) and/or serious adverse events (SAEs) | From the first infusion of YK012 until 28 Days after end of treatment
  An AE is defined as any untoward medical event that occurs after a subject receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the investigational drug.
  An SAE refers to an untoward medical occurrence such as death, life-threatening event, permanent or serious disability or loss of function, need for hospitalization or prolongation of hospitalization after the subject receives the investigational drug, and congenital abnormalities or birth defects.
The incidence and profile of dose-limiting toxicity (DLT) | 28 days after the first dose
  The toxicities occurring within 28 days (i.e., DLT observation period) after the first dose will be defined as DLTs in the discretion of the investigator as possibly, probably, or definitely related to the IMP (Investigational Medicinal Product).
The maximum tolerated dose and/or the recommended dose for further clinical trial | 28 days after the first dose
  The MTD will be determined based on the occurrence rate of the DLT. The MTD is defined as the highest dose in which 1/6 or less subjects experience a DLT.

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) after administration | 12 weeks
  Assess the AUC after treatment with YK012
Maximum concentration (Cmax) after administration | 12 weeks
  Assess the Cmax after treatment with YK012
Time to maximum concentration (Tmax) after administration | 12 weeks
  Assess the Tmax after treatment with YK012
Terminal elimination half-life (T1/2) after administration | 12 weeks
  Assess the terminal elimination half-life (T1/2) after treatment with YK012
Percentage of participants with anti-drug antibodies (ADA) | 24 weeks
  Assess the percentage of participants with ADA after treatment with YK012
Tumor objective response rate (ORR) | 24 weeks
  Assess the overall response rate (ORR) after treatment with YK012
Duration of response (DOR) | 24 weeks
  Assess the duration of response (DOR) after treatment with YK012
Anti-lymphoma activity by progression-free survival (PFS) | 24 weeks
  Assess the progression-free survival (PFS) after treatment with YK012
Number of B cells and T cells in peripheral blood after administration | 12 weeks
  Assess the number of B cells and T cells in peripheral blood after treatment with YK012
Level of cytokines in peripheral blood after administration | 12 weeks
  The activation of immune effector cells was monitored by the measurement of peripheral blood cytokine levels including interferon gamma (IFN-ɣ), interleukin (IL)-2, IL-4, IL-6, IL-8, IL-10, IL-12 and tumor necrosis factor-alpha (TNF-α) .

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China